CLINICAL TRIAL: NCT01597986
Title: A Phase 1, Open Label Study to Evaluate the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of a Single Dose Oral Contraceptive Containing Ethinyl Estradiol and Norethindrone
Brief Title: Drug Interaction Study of Isavuconazole and Oral Contraceptive Containing Ethinyl Estradiol and Norethindrone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0031
Record Dates: First submitted 2012-05-07; First posted 2012-05-15 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Pharmacokinetics of Isavuconazole; Pharmacokinetics of Ethinyl Estradiol and Norethindrone; Healthy Volunteers
Keywords: isavuconazole; ethinyl estradiol; norethindrone; contraceptive; Healthy Volunteers; BAL8557; BAL4815
MeSH Terms: interventions — isavuconazole; Contraceptives, Oral; Ethinyl Estradiol; Norethindrone; Norinyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isavuconazole and oral contraceptive (Experimental): Arm description(as needed): Subjects receive single dose of oral contraceptive consisting of ethinyl estradiol and norethindrone on Days 1 and 13 and oral doses of isavuconazole every 8 hours on Days 9 and 10 followed by a once a day dose in the mornings on Days 11 through 16.
  Interventions: Drug: isavuconazole; Drug: Oral Contraceptive (ethinyl estradiol / norethindrone)

INTERVENTIONS:
Drug: isavuconazole — oral
  Other Names: BAL8557; BAL4815
Drug: Oral Contraceptive (ethinyl estradiol / norethindrone) — contraceptive pill consisting of ethinyl estradiol and norethindrone
  Other Names: Ortho-Novum

SUMMARY:
The purpose of this study is to assess the effect of multiple doses of isavuconazole on the pharmacokinetics (PK) of a single dose of contraceptive in healthy post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and has a body mass index (BMI) of 18 to 32 kg/m2, inclusive
* Results for aspartate aminotransferase (AST), alanine aminotransferase (ALT), and total bilirubim must not be above upper limit of normal range
* The subject must be postmenopausal, defined as at least 2 years since the last regular menstrual cycle and have follicle stimulating hormone (FSH) > 30 IU/L

Exclusion Criteria:

* The subject has had treatment with hormone replacement therapy within 3 months prior to Day -1
* The subject has a history of adverse events with taking oral contraceptives or hormone replacement therapy
* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes)
* The subject has a positive result for hepatitis C antibodies or hepatitis B surface antigen at Screening or is known to be positive for human immunodeficiency virus (HIV)
* The subject has a known or suspected allergy to any of the components of the trial products or the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods (as judged by the investigator), or a history of severe anaphylactic reactions
* The subject is a smoker (any use of tobacco or nicotine containing products) within 6 months prior to Screening
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Day -1, or over-the-counter medications within 1 week prior to Day -1, with the exception of acetaminophen up to 2 g/day
* The subject has a recent history (within the last 2 years) of drug or alcohol abuse, as defined by the investigator, or a positive drug and/or alcohol screen

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) variables for ethinyl estradiol and norethindrone (in plasma): AUCinf , AUClast, and Cmax | For Days 1 and 13: predose and 12 times post dose; for Days 2, 3, 4, 5, 14, 15, 16, and 17: one time each day
  AUC from time 0 extrapolated to infinity (AUCinf), Area under the curve (AUC) from time of dosing to last quantifiable concentration (AUClast ), and maximum concentration (Cmax)

SECONDARY OUTCOMES:
PK variable for ethinyl estradiol and norethindrone (in plasma): tmax , t1/2 , Vz /F, and CL/F | For Days 1 and 13: pre-dose and 12 times post dose; for Days 2, 3, 4, 5, 14, 15, 16, and 17: one time each day
  Time to attain Cmax (tmax) , apparent terminal elimination half-life (t1/2 ), apparent volume of distribution (Vz /F), apparent body clearance after oral dosing (CL/F)
PK variable for isavuconazole (in plasma): Ctrough | For Day 11: predose; for Days 12 and 13: predose and 12 times post dose; for Day 14 and 15: predose; and for Day 16: predose and 24 hours post dose
  trough concentration (Ctrough)
PK variable for isavuconazole (in plasma): AUCtau, Cmax, and tmax | For Days 12 and 13: predose and 12 times post dose
  Area under the concentration-time curve during the time interval between consecutive dosing (AUCtau)
Safety assessed by recording adverse events, laboratory assessments, vital signs, electrocardiograms (ECGs) | Day 1 through Day 24 ± 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States